CLINICAL TRIAL: NCT06155981
Title: Coke Zero for the Zero: A Study Examining the Effect of Coke Zero Consumption on Night Call Inpatient Course and Mortality
Brief Title: Coca-Cola Zero (®) Consumption on Night-call Inpatient Course and Mortality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Kwan Yu Heng, Principle Investigator, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DukeNushssrkyh-01
Record Dates: First submitted 2023-11-18; First posted 2023-12-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mortality
Keywords: Coke Zero; Night-call Staffs; Inpatient Admission; Inpatient Course; Inpatient Mortality
MeSH Terms: interventions — Coke

STUDY DESIGN:
Intervention Model Description: Two groups of night-call staffs will be receiving different interventions.
Who Masked: Participant
Masking Description: Participants will not be aware of the type of drink they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coke Zero Arm (Experimental): The participant will be given a Coke Zero before each night-call duty for consumption.
  Interventions: Other: Coke Zero
- Coke Arm (Active Comparator): The participant will be given a Coke before each night-call duty for consumption.
  Interventions: Other: Coke

INTERVENTIONS:
Other: Coke Zero — Coca-Cola Zero Sugar drink will be given.
  Arms: Coke Zero Arm
Other: Coke — Coca-Cola drink will be given.
  Arms: Coke Arm

SUMMARY:
The purpose of this study is to determine the effect of coke zero consumption by night-call staffs on inpatient admission and mortality, and total sleep duration during the night-call duty. Coke Zero is a soft drink that is widely popular within the medical community, carrying the meaning of "zero", which to some, signifies the minimal level of morbidity and mortality that will occupy the on-call the night staffs.

DETAILED DESCRIPTION:
Previous studies have demonstrated that superstitions among the medical community have been prevalent and staffs regularly engaged in conforming to the superstitions because of their associations with workload, inpatient admissions and mortality. As such, the current study aims to evaluate whether the consumption of Coke Zero has an effects on patient admissions and mortality and the eventfulness of the night-call duties.

ELIGIBILITY:
Inclusion Criteria:

• Doctors on the night-call roster at Singapore General Hospital

Exclusion Criteria

• Other allied health professionals or medical students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Inpatient Mortality | The designated night-call doctor's shift from 5PM to 8AM the next day
  For patients assigned under the designated night-call doctor's care
Inpatient general ward admission | The designated night-call doctor's shift from 5PM to 8AM the next day
  For patients assigned under the designated night-call doctor's care
Inpatient High Dependency/Intensive Care Unit Admission | The designated night-call doctor's shift from 5PM to 8AM the next day
  For patients assigned under the designated night-call doctor's care

SECONDARY OUTCOMES:
Hours of sleep during the night-call | The designated night-call doctor's shift from 5PM to 8AM the next day
  For the designated night-call doctor's care
Hours of shift during the night-call | The designated night-call doctor's shift from 5PM to 8AM the next day
  For the designated night-call doctor's care
Number of steps walked by the night-call staff during the night-call | The designated night-call doctor's shift from 5PM to 8AM the next day
  For the designated night-call doctor's care
Level of alertness of the night-call staff after the night-call | The designated night-call doctor's shift from 5PM to 8AM the next day
  Measured using the Karolinska Sleepiness Scale and the Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yu Heng Kwan, MD, PhD, Principal Investigator — SingHealth Internal Medicine Residency
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD to other researchers.

REFERENCES:
- [Background] Tan MH, Lee Z, Ng B, Sim ES, Chua YY, Tien M, Ooi CJ. The Tao of bao: a randomised controlled trial examining the effect of steamed bun consumption on night-call inpatient course and mortality. Ann Acad Med Singap. 2008 Mar;37(3):255-3. PMID 18392313